CLINICAL TRIAL: NCT06524323
Title: A Randomized, Double-blinded, Self-controlled Clinical Study of Intralesional Injection of 5-fluorouracil Plus Triamcinolone for the Treatment of Refractory Nodular Prurigo
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Xiaoyong Man, Director, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-0042
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Nodular Prurigo
Keywords: nodular prurigo; 5-fluorouracil
MeSH Terms: interventions — Fluorouracil; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control side (Other): Intralesional injection of triamcinolone acetonide alone
  Interventions: Drug: Triamcinolone Acetonide
- Experimental side (Experimental): Intralesional injection of 5-fluorouracil plus triamcinolone acetonide
  Interventions: Drug: 5-fluorouracil Injection

INTERVENTIONS:
Drug: 5-fluorouracil Injection — The mixture contains 2mL of triamcinolone acetonide injection and 4mL of 5-fluorouracil injection, which is diluted with saline to 10mL.
  Arms: Experimental side
Drug: Triamcinolone Acetonide — The mixture contains 2mL of triamcinolone acetonide injection which is diluted with saline to 10mL.
  Arms: Control side

SUMMARY:
Nodular pruritus is a chronic inflammatory skin disease manifested as individual or multiple highly keratotic nodules with severe itching. The goal of this clinical trial is to compare the efficacy and safety of treating refractory nodular pruritus with intralesional injections of 5-fluorouracil alone or 5-fluorouracil plus triamcinolone acetonide.

DETAILED DESCRIPTION:
The study is a single-center, randomized, double-blinded, self-controlled clinical trial and is expected to enroll 60 patients. The trial is set up with a self-control design, comparing the two treated sides on the arms or legs with 1:1 interindividual randomization (right side: triamcinolone acetonide-alone; left side: 5-fluorouracil plus triamcinolone acetonide; or the other way round). Patients who meet all the inclusion criteria and do not meet any of the exclusion criteria are randomly enrolled and receive trial medication treatment. All enrolled patients with receive intralesional injections of the trial medication once every 4 weeks for a total of 12 weeks. For the first 4 weeks after the initial dose, follow-up visits are scheduled every 2 weeks; from weeks 5 to 12, follow-up visits are scheduled every 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 1) Fully understand and voluntarily sign an informed consent form for this experiment;
* 2) When signing the informed consent form, the age of male or female participants is ≥ 18 years old and ≤ 70 years old;
* 3) During the screening of subjects, the onset time of nodular prurigo was at least 6 months, and it met the diagnostic criteria for nodular prurigo;
* 4) Within the 12 weeks before screening, no intralesional injection of triamcinolone acetonide or 5-FU combined with triamcinolone acetonide treatment was received;
* 5) Within the specified time window before screening, there is a clear medical history showing that patients who have received any of the following treatment regimens can partially alleviate nodular prurigo but have not been completely cleared:

  1. Continuous use of systemic therapies such as antihistamines, antiepileptic drugs (gabapentin, pregabalin, etc.), glucocorticoids, or immunosuppressants (methotrexate, cyclosporine, thalidomide, etc.) for the first 4 weeks before screening;
  2. Continuous use of small molecule inhibitors (including tofacitinib/tofacitinib, baritinib/baritinib, Upadacitinib/Upatinib, Abrocitinib/Abrocitinib, ruxolitinib/Lucetinib, filgotinib/Figetinib, lestaurtinib/letatinib, pacritinib/parkatinib, Delgocitinib, SHR0302, etc.) for the first 4 weeks before screening;
  3. Continuous use of biologics (including monoclonal antibodies targeting IL-4, IL-13, IL-31, IgE, etc.) for the first 8 weeks before screening;
  4. Continuous use of phototherapy (such as UVB, PUVA, etc.) for the first 4 weeks before screening;
* 6) From the start of screening until the end of the visit, the subject can only continue to use moisturizers and the treatment regimens listed in the Inclusion Criteria 5;
* 7) Multiple symmetrically distributed nodules (10-12 nodules on one side) were observed in the trunk and limbs during subject screening;
* 8) During the subject screening, the Pruritus Numerical Rating Scale (NRS) score was ≥ 4 points;
* 9) For women with reproductive ability and all male subjects, abstinence or contraception must be maintained during the trial period and for 6 months after discontinuation of the trial drug:
* 10) The subjects can communicate well and agree to comply with the study and follow-up procedures.

Exclusion Criteria:

* 1) Have other inflammatory skin diseases (such as psoriasis), as well as any abnormal skin changes that may affect the evaluation of treatment response for nodular prurigo;
* 2) Known or suspected allergy to 5-fluorouracil and its analogs;
* 3) Have received aspirin drugs within the first week before screening and need to be taken for a long time, and should not be discontinued;
* 4) Within the specified time window before the first administration, individuals with the following infection status:

  1. Patients with active tuberculosis (TB), latent untreated TB, or a history of TB or non-tuberculous mycobacterium infection with potential incomplete treatment within 48 weeks before screening, or patients with TB screening indicating latent TB infection;
  2. The following infections that are active and uncontrolled during screening: HIV positive, active syphilis, HBsAg positive for hepatitis B with HBV-DNA detection values exceeding the lower limit of quantification, positive anti-HCV antibodies or HCV-RNA positive for hepatitis C;
  3. Screening for bacterial, viral, mycoplasma, parasitic, protozoan, or fungal infections with any clinical symptoms within the first two weeks that require systemic anti-infection treatment, or screening for individuals with active lung infections indicated by chest imaging examination;
  4. Screening for individuals with a history of herpes simplex virus or varicella-zoster virus infection within the first 4 weeks, or those with superficial skin infections that require treatment within the first week but have not recovered;
* 5) Individuals with the following serious chronic or acute diseases that have not been controlled:

  1. Have a clear history of arterial or venous thromboembolism within the first 12 weeks of randomization, or have a high-risk state that requires long-term use of anticoagulants to prevent thrombosis;
  2. Individuals with severe heart disease within the first 12 weeks of randomization, including myocardial infarction, heart failure (grade III or IV according to the NYHA classification), history of unstable angina, or third-degree atrioventricular block and other life-threatening arrhythmias;
  3. Individuals who have experienced severe trauma or major surgery within the first 4 weeks of randomization;
  4. Serious neurological disorders were present during screening, including acute cerebrovascular diseases within the first 6 months of randomization, previous seizures within the first 4 weeks of randomization or the need for continuous anti-epileptic drug treatment, known or suspected demyelinating neurological disorders during screening, peripheral neuropathy with CTCAE V5.0 ≥ 2, and any significant neurological dysfunction remaining;
  5. During screening, there were severe mental illness patients, including any severe/unstable mental/psychological illness or somatic illness/symptoms, as well as recent or current suicidal thoughts or behaviors, as well as other researchers who believed they would pose an unacceptable risk to participants in the study, except for those with mild emotional disorders caused by nodular prurigo who do not require antipsychotic or sedative maintenance therapy;
  6. When screening, individuals with known or suspected immunodeficiency diseases, first-degree relatives with hereditary immunodeficiency diseases, or those who have received organ transplants that require sustained immunosuppression;
  7. There is known or suspected leukopenia during screening;
  8. Individuals with a known or suspected history of thrombocytopenia, coagulation disorders, or platelet dysfunction during screening;
  9. Have other serious and uncontrolled diseases, including severe lung, liver, kidney, endocrine and metabolic, lymphatic system, autoimmune and connective tissue diseases, etc;
* 6) Have the following events within the specified time window before the first administration of the investigational drug:

  1. Individuals with a history of drug abuse, alcohol abuse, or addiction, including those who frequently (>3 times per week) use sedatives, sleeping pills, or tranquilizers;
  2. Individuals who have received any clinical trial treatment of drugs or medical devices within the first 4 weeks of randomization;
  3. When screening, there is a clear plan to undergo major surgeries during the study period, or significant changes in work and life status that may affect compliance with the study;
* 7) During screening or baseline visits, laboratory tests did not meet the following criteria:

  1. Blood routine: WBC count ≥ lower limit of normal (LLN), neutrophil count ≥ LLN, lymphocyte count ≥ LLN, platelet count ≥ 100 × 109/L, hemoglobin ≥ 100g/L;
  2. Liver function indicators: ALT<2.0 x ULN, AST<2.0 x ULN, total bilirubin<1.5 x ULN;
  3. Renal function indicators: glomerular filtration rate (eGFR) ≥ 60 ml/min/1.73 m2;
  4. Blood glucose: Fasting blood glucose<8.9mmol/L (allowed to be controlled by hypoglycemic drugs);
  5. Blood pressure: systolic blood pressure<160mmHg and/or diastolic blood pressure<100mmHg (allowed to be controlled by no more than two antihypertensive drugs);
  6. Coagulation function indicators: PT<1.5 x ULN, APTT<1.5 x ULN, INR<1.5;
  7. 12 lead electrocardiogram QTc<480ms, cardiac ultrasound LVEF ≥ lower limit of normal value;
* 8) The researchers believe that any other subjects who are unsuitable to participate in this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Clearance rate | Week 12 after administration
  The proportion of subjects with a clearance rate of ≥ 90%
NRS score | Week 12 after administration
  The proportion of subjects whose NRS score improved by ≥ 4 points from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No